CLINICAL TRIAL: NCT02042404
Title: The EarLens System Long Term Safety and Efficacy Definitive Multi-Center Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EarLens Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EarLens CRP00004
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Hearing Impairment
Keywords: Hearing impairment; Hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mild to severe hearing impairment (Experimental): Sound amplification provided via the EarLens System assistive hearing device.
  Interventions: Device: Sound amplification provided via EarLens System.

INTERVENTIONS:
Device: Sound amplification provided via EarLens System. — The EarLens System has two primary components: 1) an external Behind the Ear (BTE) Sound Processing Unit, and 2) a Tympanic Membrane Transducer (TM Transducer). In this system, light is used to wirelessly transmit both signal and power from the BTE Sound Processor to the TM Transducer. The BTE is designed to be able to be removed, reprogrammed, and have the battery recharged as needed, similar to a BTE for an air conduction hearing aid. The removable TM Transducer is customized for each patient, is placed and removed by a physician in an office visit procedure, and is designed to reside in the ear in a safe and stable manner for long periods of time.

SUMMARY:
The EarLens System is an assistive hearing device that is intended to provide amplification for the treatment of patients with sensorineural hearing impairment. The purpose of this multi-center definitive study is to assess the safety and efficacy of the EarLens System for subjects with bilateral mild to severe sensorineural hearing impairments wearing the fully activated system in their daily lives for a 4 month period of time. This study is designed to support US and International marketing applications to commercialize the EarLens System. The main efficacy hypothesis is that the EarLens System will be shown to improve speech understanding in quiet.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years
* Mild to severe hearing impairment between 125 to 4000 Hz
* No significant conductive hearing impairment
* Able and willing to commit to travel and time demands of the study

Exclusion Criteria:

* Must not have known or active medical issues that would preclude having a device including:

  1. an abnormal tympanic membrane
  2. an abnormal middle ear or history of prior middle ear surgery other than tympanostomy tubes
  3. an ear canal anatomy that prevents physicians from seeing adequate amount of the tympanic membrane
* Must not have other known or active medical issues including:

  1. history of chronic and recurrent ear infections in the past 24 mouths
  2. history of dizziness and/or vertigo in the past 24 months
  3. taking medications/treatments with known ototoxic effects
  4. a rapidly progressive or fluctuating hearing impairment
  5. having been diagnosed with having a compromised immune system
* Must not fit the definition of a vulnerable subject, as per FDA regulations 21 CFR Parts 50 and 56
* Must not have an ear canal anatomy that preclude manufacture of the device as determined by EarLens manufacturing personnel

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Gantz, M.D., Principal Investigator — University of Iowa Dept of Otolaryngology--Head and Neck Surgery University of Iowa Hospitals and Clinics; Sunil Puria, Ph.D., Study Chair — EarLens Corp.
Locations (3):
- United States (3):
  - EarLens Corporation, Menlo Park, California
  - Camino Ear Nose and Throat Clinic, San Jose, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa

REFERENCES:
- [Background] Fay JP, Perkins R, Levy SC, Nilsson M, Puria S. Preliminary evaluation of a light-based contact hearing device for the hearing impaired. Otol Neurotol. 2013 Jul;34(5):912-21. doi: 10.1097/MAO.0b013e31827de4b1. PMID 23524632
- [Derived] Arbogast TL, Moore BCJ, Puria S, Dundas D, Brimacombe J, Edwards B, Carr Levy S. Achieved Gain and Subjective Outcomes for a Wide-Bandwidth Contact Hearing Aid Fitted Using CAM2. Ear Hear. 2019 May/Jun;40(3):741-756. doi: 10.1097/AUD.0000000000000661. PMID 30300158
- See also: EarLens Corporation website — http://www.earlenscorp.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Flyers approved by WIRB for subject recruitment. Also referrals from local audiology clinics and otologists.
Pre-assignment Details: The first five (5) enrolled will be part of a pilot phase of the study to work out the process flow and training of the centers and participants, called "Roll-in Cohort."
Groups:
- Primary Cohort: Mild to Severe Hearing Impairment: Sound amplification provided via the EarLens System assistive hearing device.
  Sound amplification provided via EarLens System.: The EarLens System has two primary components: 1) an external Behind the Ear (BTE) Sound Processing Unit, and 2) a Tympanic Membrane Transducer (TM Transducer). In this system, light is used to wirelessly transmit both signal and power from the BTE Sound Processor to the TM Transducer. The BTE is designed to be able to be removed, reprogrammed, and have the battery recharged as needed, similar to a BTE for an air conduction hearing aid. The removable TM Transducer is customized for each patient, is placed and removed by a physician in an office visit procedure, and is designed to reside in the ear in a safe and stable manner for long periods of time.
- Roll-in Cohort: Mild to Severe Hearing Impairment: Roll-in Cohort are evaluated for safety only, and are not included in efficacy endpoint evaluation.
Period: Overall Study
Arm/Group | Primary Cohort: Mild to Severe Hearing Impairment | Roll-in Cohort: Mild to Severe Hearing Impairment
Started | 43 (Enrollment was stopped after 43 were enrolled, had approval to enroll 45 primary cohort subjects) | 5
Completed | 38 (39 subjects completed 30 days evaluation. 38 subjects completed 120 days evaluation.) | 5
Not Completed | 5 | 0
Not completed — Death | 1 | 0
Not completed — Unrelated Adverse Event | 3 | 0
Not completed — Inability to meet time requirements | 1 | 0

BASELINE CHARACTERISTICS:
Population: Both Primary Cohort and Roll-in Cohorts combined in Demographic Report
Groups:
- Mild to Severe Hearing Impairment: Subjects wearing the Earlens System in their daily lives.
Arm/Group | Mild to Severe Hearing Impairment
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Aided Word Recognition Scores (WRS) When Compared to the Baseline Unaided Condition.
Description: Change in mean aided Word Recognition Scores (WRS) when compared to the baseline unaided condition. WRS will be measured using 50-word NU-6 (Northwestern University Auditory Test No.6) recorded materials, presented at 45 dB Hearing Level on a per-ear basis with the test ear isolated for measurement and the results, expressed as a percentage of words correct, averaged across the two ears for each subject. All subject data will then be averaged to obtain the means. The baseline unaided measurements will occur prior to device placement, and the aided condition will be measured at least 30 days post device placement.
Time Frame: Baseline and 30 days
Population: 39 subjects available for analysis between enrollment/treatment and 30 day measurement.
Measure: Mean (Standard Deviation); unit: percentage of words correctly identified
Arm/Group | Primary Cohort: Mild to Severe Hearing Impairment | Roll-in Cohort: Mild to Severe Hearing Impairment
Number analyzed (Participants) | 39 | 0
percentage of words correctly identified | 37.6 (24.6) |
Statistical Analysis 1: Comparison: Primary Cohort: Mild to Severe Hearing Impairment; Test type: Superiority or Other; p < 0.0001, repeated measures ANOVA

2. Primary Outcome: Audiometric Safety as Shown by no Hearing Change Pre and Post Treatment
Description: The unaided air conduction hearing thresholds will be measured for each individual ear twice before device placement at Visit #1 and averaged to obtain the baseline unaided air conduction hearing thresholds, and the post wear unaided air conduction hearing thresholds will be measured after device removal at Visit #5. A PTA4 (Pure Tone Average at 4 frequencies; 500, 1000, 2000, and 4000 Hz) will be computed both for baseline unaided hearing pre-placement and unaided hearing post-removal for each ear, then averaged across both ears for each subject . A determination of "No Hearing Change" for the subject population will be made if the calculated Hearing Changes of the subject population are 10 dB or less.
Time Frame: Baseline and 120 days
Population: 43 subjects available for analysis between enrollment/treatment and 120 day measurement.
Measure: Mean (Standard Deviation); unit: dB difference in Unaided Hearing
Groups:
- Mild to Severe Hearing Impairment: Both Primary Cohort and Roll-in Cohorts are combined for safety analysis.
Arm/Group | Mild to Severe Hearing Impairment
Number analyzed (Participants) | 43
dB difference in Unaided Hearing | -0.3983 (2.9822)
Statistical Analysis 1: Comparison: Mild to Severe Hearing Impairment; Test type: Superiority or Other; p < 0.0001, repeated measures ANOVA

3. Secondary Outcome: Functional Gain Over the Frequency Range From 2000 to 10,000 Hz
Description: 10 dB (decibel) change in the averaged pure tone thresholds for the subject population over the frequency range from 2000 to 10,000 Hz (2000, 3000, 4000, 6000, 8000, 9000 and 10,000 Hz). Measurement to be used in analysis are the baseline unaided soundfield thresholds measured prior to device placement and the aided soundfield thresholds measured at least 30 days post placement. Analysis includes calculation of the unaided soundfield thresholds minus aided soundfield thresholds.
Time Frame: Baseline and 30 days
Population: 39 subjects available for analysis between enrollment/treatment and 30 day measurement.
Measure: Mean (Standard Deviation); unit: dB difference in Soundfield Hearing
Arm/Group | Primary Cohort: Mild to Severe Hearing Impairment | Roll-in Cohort: Mild to Severe Hearing Impairment
Number analyzed (Participants) | 39 | 0
dB difference in Soundfield Hearing | 30.4819 (10.2504) |
Statistical Analysis 1: Comparison: Primary Cohort: Mild to Severe Hearing Impairment; Test type: Superiority or Other; p < 0.0001, repeated measures ANOVA

4. Secondary Outcome: Change in Aided HINT 90 Speech Reception Thresholds (SRTs) When Compared to the Baseline Unaided Condition.
Description: Change in aided HINT 90 speech reception thresholds (SRTs) when compared to the baseline unaided condition. SRTs will be measured using HINT materials with the signal (speech level presented from 0 degrees) adapted relative to the noise (presented from 90 degrees held fixed at 60 dB SPL) to determine the signal-to-noise ratio for reporting the whole sentence correct 50% of the time (Nilsson et al., 1994). An improvement in HINT score is indicated as a negative (-) dB value change. A more negative value indicating an improvement of understanding speech and noise. An improvement of -1dB is equivalent to a 10% improvement in understanding speech and noise and is likely of clinical benefit. HINT 90 will be measured twice and averaged to obtain the per subject HINT SRT. All subject data will be averaged to obtain the means. Analysis includes calculation of the unaided measurements (before device placement) minus the aided measurements.
Time Frame: Baseline and 30 days
Population: 39 subjects available for analysis between enrollment/treatment and 30 day measurement.
Measure: Mean (Standard Deviation); unit: dB difference in HINT scores
Arm/Group | Primary Cohort: Mild to Severe Hearing Impairment | Roll-in Cohort: Mild to Severe Hearing Impairment
Number analyzed (Participants) | 39 | 0
dB difference in HINT scores | 0.7542 (4.2207) |
Statistical Analysis 1: Comparison: Primary Cohort: Mild to Severe Hearing Impairment; Test type: Superiority or Other; p = 0.0281, repeated measures ANOVA

5. Other Pre Specified Outcome: Determine the Incidence of Serious Device- and Procedure-related Adverse Events.
Description: The analysis of the incidence of serious device- and procedure-related adverse events through the study period. All adverse events will be recorded on case report forms and determinations will be made as to the whether the events are related to the investigational device.
Time Frame: 120 days
Population: Both Primary Cohort and Roll-in Cohort were included in all safety analyses.
Measure: Number; unit: serious device- or procedure-related AEs
Arm/Group | Mild to Severe Hearing Impairment
Number analyzed (Participants) | 48
serious device- or procedure-related AEs | 0

ADVERSE EVENTS:
Arm/Group | Mild to Severe Hearing Impairment
Serious Adverse Events (participants affected / at risk) | 5/48
Other Adverse Events (participants affected / at risk) | 25/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild to Severe Hearing Impairment (N=48)
Altered mental status (Psychiatric disorders) | 1 (1) — Not device related.
Hospitalized for bike accident (Injury, poisoning and procedural complications) | 1 (1) — Not device related.
Drug overdose leading to death (Psychiatric disorders) | 1 (1) — Not device related.
Bacterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not device related.
Hospitalized for heart issues (Cardiac disorders) | 1 (1) — Not device related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild to Severe Hearing Impairment (N=48)
Abrasion/Blood blister in the ear canal (Ear and labyrinth disorders) | 13 (17) — Device related, anticipated, mild, all resolved.
Abrasion/Blood/Blister on tympanic membrane (Ear and labyrinth disorders) | 2 (2) — Device related, anticipated, mild, all resolved.
Ear discomfort/pain (Ear and labyrinth disorders) | 5 (5) — Device related, anticipated, mild/moderate, all resolved.
Ear tip, other: swelling, itching (Ear and labyrinth disorders) | 2 (2) — Device related, anticipated, mild/moderate, all resolved.
Inflammation/Granulation tissue on tympanic membrane (Ear and labyrinth disorders) | 3 (3) — Device related, anticipated, mild, all resolved.
Pain upon eructation/ valsalva (Ear and labyrinth disorders) | 1 (1) — Device related, anticipated, mild, all resolved.
Pressure sensation of device on tympanic membrane (Ear and labyrinth disorders) | 1 (1) — Device related, anticipated, mild, ongoing as subject continues to wear the device..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No